CLINICAL TRIAL: NCT01904877
Title: Multi-component HIV Intervention Packages for Chinese Men Who Have Sex With Men -Test, Link and Care (TLC) Version 1.0 Dated 10/15/12
Brief Title: Multi-component HIV Intervention Packages for Chinese Men Who Have Sex With Men -Test, Link and Care (TLC)
Acronym: MP3
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Responsible Party: Sponsor
Other Study IDs: 11914
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: HIV/AIDS
Keywords: HIV testing; linkage; care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — HIV RNA will be extracted from plasma and the HIV PR and RT genes will be amplified by a one-step RT-PCR using TaKaRa One Step RNA PCR Kit . The quality of sequences will be evaluated using Sequence Scanner v1.0, and the sequences will be cleaned and assembled by Sequencher (Gene Codes Corporation, Ann Arbor, MI,USA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV testing: Enhancing HIV testing: By partnering with the local CDC and the gay community, we will use SMS-I intervention by cell phones, web advertisement, community outreach, and peer referral strategies to recruit MSM in Beijing City for receiving HIV testing.
  Interventions: Behavioral: Enhancing HIV testing
- Phase II: 367 HIV positive MSM: * Linking to care:
  * Providing enhanced HIV care.

INTERVENTIONS:
Behavioral: Enhancing HIV testing — SMS-I intervention by cell phones, web advertisement, community outreach, and peer referral strategies to recruit MSM in Beijing City for receiving HIV testing
  Other Names: Phase I
  Groups: HIV testing

SUMMARY:
1. The number of MSM who are tested for HIV in the 4 study clinics over 12 months will increase compared with historical data from the same 4 clinics over the past 12 months prior to the intervention.
2. Persons diagnosed with HIV over the duration of 12 months will have higher CD4 counts at diagnosis than persons diagnosed with HIV over the past 12 months prior to the intervention

ELIGIBILITY:
Inclusion Criteria:• Men who had sex with another man in the last 12 months based on self-reporting (sex can be defined as oral, anal, or mutual masturbation)(including transgendered women)（including transgendered women）;

* Aged 18 years or older;
* Living and/or working in the defined districts of municipal Beijing;
* Able and willing to adequately grant informed consent. For the purposes of this activity participants must consent to questionnaire surveys, receipt of phone messages, and serological testing;
* Having not previously participated in HIV testing in this study.

Besides these criteria, additional criteria for the HIV Linkage and Care pilot Research Clinical Trial are:

* Men who are being identified as HIV positive during the testing campaign in Phase I of the study;
* No plan to leave Beijing in the next 12 months.
* Willing to comply with study procedures.
* Having a cell phone and willing to receive study related SMS texts

Exclusion Criteria:

Having previously been found to be HIV positive based on self-reporting during eligibility screening;

* Serious psychological disturbance or cognitive impairment interfering with the participant's ability to comply with the study visit schedule and procedures, as judged by the local study clinician;
* Any other medical or psychiatric condition that, in the opinion of the investigator, would make participation in the study unsafe, or otherwise interfere substantially with the study objectives or interpretation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects selected are living or working in Beijing China
Sampling Method: Probability Sample
Enrollment: 3760 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
(Primary) phase I: The number of MSM who are tested for HIV in 4 study clinics over 12 months will increase significantly compared with historical data from the same 4 clinics over the past 12 months prior to the intervention | 12 months
  The effect of intervention on the monthly number of MSM who receive HIV testing prior to and after intervention at 4 clinics will be evaluated using a generalized estimating equation (GEE) model with robust variance estimates to account for correlation in outcomes within a clinic
Phase II: A higher proportion of participants in the intervention arm will obtain their CD4 results and ART eligibility assessment in a CDC clinic within 1 month of being diagnosed with HIV than in the comparison arm experienced a local standard of care. | 1 month
  The proportion of participants randomized to the intervention arm who obtain their CD4 count results within 1 month of randomization will be compared to the same proportion in the comparison arm using logistic regression. The primary analysis will adjust for the following baseline covariates: clinic, CD4 count, ART eligibility, self-reported drug abuse, self-reported alcohol abuse, and age.

SECONDARY OUTCOMES:
Phase I: Persons diagnosed with HIV over the duration of 12 months will have higher CD4 counts at diagnosis than persons diagnosed with HIV over the past 12 months prior to the intervention. | 12 month
  We will compare the distribution of CD4 counts immediately after HIV diagnosis for all MSM diagnosed with HIV at one of the 4 clinics for the 12 months during the intervention period versus the 12 months prior to the intervention using a Wilcoxon rank sum test
Phase II:A higher proportion of ART eligible participants in the intervention arm will receive their first HIV medical care within 3 months of diagnosis than in the comparison arm. | 12 months
  A logistic regression analysis will be performed to assess the association between intervention and timely receipt of first HIV medical care among those who are ART eligible (CD4<350). The analysis will adjust for the following baseline covariates: clinic, CD4 count, self-reported drug abuse, self-reported alcohol abuse, and age.

OTHER OUTCOMES:
Phase II: A higher proportion of participants in the intervention arm will obtain their CD4 results and ART eligibility assessment in a CDC clinic within 1 month of being diagnosed with HIV than in the comparison arm experienced a local standard of care. | 36 months
  To evaluate the efficacy of interactive SMS-II with peer education/counseling intervention for reducing risky sexual behaviors among HIV-infected Chinese MSM over the first year of HIV-care

CONTACTS AND LOCATIONS:
Overall Officials: Sten H Vermund, MD,PhD, Study Chair — Vanderbilt Institue for Global Health; Han-Zhu Qian, MD,PhD, Study Director — Vanderbilt Institue for Global Health; Yiming Shao, MD,PhD, Study Director — Division of Immunology and Microbiology NCAIDS, China CDC

REFERENCES:
- [Derived] Liu Y, Vermund SH, Ruan Y, Liu H, Rivet Amico K, Simoni JM, Shepherd BE, Shao Y, Qian HZ. Peer counselling versus standard-of-care on reducing high-risk behaviours among newly diagnosed HIV-positive men who have sex with men in Beijing, China: a randomized intervention study. J Int AIDS Soc. 2018 Feb;21(2):e25079. doi: 10.1002/jia2.25079. PMID 29430845